CLINICAL TRIAL: NCT01019551
Title: International, Multicenter, Randomized, Non-comparative Controlled Study of Therapeutic Intensification Plus Immunomodulation in HIV-infected Patients With Long-term Viral Suppression
Brief Title: Therapeutic Intensification Plus Immunomodulation in HIV-infected Patients
Acronym: ERAMUNE-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Objectif Recherche Vaccins SIDA (Other)
Collaborators: Cytheris SA (Industry); Merck Sharp & Dohme LLC (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORVACS 010
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: HIV-1 Infection
Keywords: Controlled viremia; Viral reservoirs; Virus eradication; Therapeutic intensification; Immunointervention
MeSH Terms: interventions — Immunomodulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM A : ART intensification alone (Experimental): Raltegravir PO 400 mg BID Maraviroc PO 150, 300 or 600 mg BID depending on the concomitant ART regimen
  Interventions: Drug: ART Intensification
- ARM B : ART intensification + Immunomodulation (Experimental): Raltegravir PO 400 mg BID during 56 weeks Maraviroc PO 150, 300 or 600 mg BID depending on the concomitant ART regimen during 56 weeks 3 weekly injections of r-hIL-7 (CYT107) at a 20 micrograms/kg dose starting at Week 8
  Interventions: Drug: ART Intensification; Biological: Immunomodulation

INTERVENTIONS:
Drug: ART Intensification — Current ART regimen plus raltegravir and maraviroc Raltegravir : 400 mg PO BID for 56 weeks Maraviroc : 150, 300 or 600 mg PO BID depending on concomitant ART treatment, for 56 weeks
Biological: Immunomodulation — Starting at Week 8, 1 cycle of 3 injections (1 per week) of recombinant human Interleukin-7 (r-hIL-7 / CYT107) at a 20 µg/kg dose.
  Arms: ARM B : ART intensification + Immunomodulation

SUMMARY:
Viral eradication in selected HIV-infected patients is possible with intensive antiretroviral therapy plus immunomodulation

DETAILED DESCRIPTION:
The overall strategy of the ERAMUNE 01 Trial is to treat selected patients with an optimal synergistic antiretroviral regimen plus one or more immunomodulating agents. Among immunomodulating treatments the candidates include therapies from two functional classes: 1) agents that target actively replicating cells and 2) agents activating latently infected cells31.

The novelty of this approach is three-fold: first, the use of highly potent antiretroviral therapy combining drugs with different HIV enzymes targets or receptors and different penetrations in cells, with the aim to suppress virus to truly undetectable levels as measured by the most sophisticated viral quantification techniques; secondly, the addition of an immunomodulatory therapy that specifically targets viral reservoirs to this intensification strategy; and lastly, the rigorous selection of patients having already a low HIV reservoir as measured by peripheral blood HIV DNA content. To our knowledge, this type of strategy has not been implemented. We believe this strategy is feasible.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed ELISA test kit and confirmed by Western Blot at any time prior to study entry. HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test
* 18 ≤ Age ≤ 70 years
* At least 3 years of suppressive ART without any interruption (less than one month cumulative),
* ART treatment unchanged in the 3 months prior to screening
* One HIV plasma viral load (RNA) documented at least 3 years prior to entry, and at least 2 HIV plasma viral loads (RNA) documented per year thereafter
* HIV plasma viral load (RNA) ≤ 500 copies/ml at least 3 years prior to entry and HIV plasma viral load ≤ 500 copies/ml for ≥ 90% of the measures thereafter
* HIV plasma viral load (RNA) below the limit of detection for all values within the past year. Note: the assay used must have a lower limit of detection of 75 copies/ml or less
* CD4+ count ≥ 350 cells/mm3 within 60 days of entry
* 10 ≤ Proviral DNA ≤ 1000 copies/106 PBMCs within 60 days of entry
* Documented laboratory values: Haemoglobin ≥ 10 g/dl, Platelets ≥ 100,000 per microliter, Hepatic transaminases ≤ 2.5 x ULN, Creatinine clearance ≥ 50 ml/min by the Cockcroft-Gault equation
* All subjects must agree not to participate in the conception process (e.g. active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, the subject/partner must use at least two reliable forms of contraceptives (condoms, with or without spermicidal agent, a diaphragm or cervical cap with spermicide, an IUD, or hormone-based contraception), while receiving study treatment and for 6 weeks after stopping study treatment
* Ability and willingness to provide informed consent.

Exclusion Criteria:

* Sexually active men and women who will not practice at least one form of barrier birth control (male partner using condoms, female partner using condoms, other barrier contraception, etc)
* Pregnancy as documented by a urine pregnancy test, or lactating women
* Hepatitis B antigen (HBsAg) positive
* Hepatitis C virus (HCV-Ab) positive or HCV RNA detectable
* Previous use of an integrase inhibitor (ie raltegravir) or a CCR5 inhibitor (ie maraviroc, vicriviroc). Use of raltegravir for non-treatment failure indications such as intensification and toxicity switches is allowed, provided that 1) virologic suppression was maintained before, during and after raltegravir treatment and 2) the patient has not received raltegravir treatment in the 6 months prior to study entry.
* Previous immunologic therapeutic intervention (e.g. IL-2, IL-7) within the past year
* Participation in another clinical drug or device trial where the last dose of drug was within the past 30 days or an investigational medical device is currently implanted
* Diagnosis of cancer within the last 5 years (except basal cell cutaneous cancers and cutaneous KS not requiring systemic therapy)
* Co-morbid condition with an expected survival less than 12 months
* History of hypersensitivity to vaccination
* History of autoimmune disease, such as systemic lupus erythematosis (SLE) or Hashimoto's thyroiditis
* Active drug or alcohol use or dependence that, in the opinion of the center investigator, would interfere with adherence to study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Decrease from baseline in HIV proviral DNA in the PBMCs at week 56 of at least 0.5 log, as expressed as numbers of HIV DNA copies per million PBMCs | End of study

SECONDARY OUTCOMES:
Percentage of patients with undetectable HIV DNA (< 1 copy/million PBMCs) after 56 weeks | End of study
Change from baseline in HIV proviral DNA in any of the sub-compartments explored (gut lymphoid tissue), as expressed as numbers of HIV DNA copies per million mononuclear cells | From Day 0 to Week 56
Change from baseline in HIV proviral DNA in the CD4 T cell subsets, as expressed as numbers of HIV DNA copies per million CD4 T cells | From Day 0 to Week 56
Changes from baseline in HIV plasma viral load (number of copies of HIV RNA per millilitre), measured by quantitative ultrasensitive PCR | From Day 0 to Week 56
Proportion of patients without inducible HIV RNA, DNA and/or p24 | End of study
Changes from baseline in CD4 lymphocyte count | From Day 0 to Week 56
Changes in the activation and differentiation markers of the CD4 and CD8 peripheral blood T cells | End of study
Development of a mathematical model exploring the dynamics of the HIV-DNA decay | From Day 0 to Week 56
Development of a mathematical model exploring the dynamics of T cells activation (CD38) | From Day 0 to Week 56
Genetic determinants influencing HIV-1-specific immune response and HIV control | End of study
Antiretroviral drugs pharmacokinetics in the blood and rectal mucosa | From Day 0 to Week 56
Safety and tolerability of the intensified treatment regimen and immunomodulatory therapy | From Day 0 to Week 56

CONTACTS AND LOCATIONS:
Overall Officials: Christine KATLAMA, MD, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière; Steven DEEKS, MD, Study Chair — University of California, San Francisco; François LECARDONNEL, MSc, Study Director — ORVACS
Locations (5):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France
- San Raffaele Scientific Institute, Milan, Italy
- Spain (2):
  - Fundacio Irsicaixa, Badalona
  - University Hospital Clinic of Barcelona, Barcelona
- Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Background] Murphy RL, Autran B, Katlama C, Brucker G, Debre P, Calvez V, Clotet B, Clumeck N, Costagliola D, Deeks SG, Dorrell L, Gatell J, Haase A, Klein M, Lazzarin A, McMichael AJ, Papagno L, Schacker TW, Wain-Hobson S, Walker BD, Youle M. A step ahead on the HIV collaboratory. Science. 2009 Jun 5;324(5932):1264-5. doi: 10.1126/science.324_1264b. No abstract available. PMID 19498149
- [Background] Lewin SR, Rouzioux C. HIV cure and eradication: how will we get from the laboratory to effective clinical trials? AIDS. 2011 Apr 24;25(7):885-97. doi: 10.1097/QAD.0b013e3283467041. PMID 21422987
- [Background] Lafeuillade A. Eliminating the HIV reservoir. Curr HIV/AIDS Rep. 2012 Jun;9(2):121-31. doi: 10.1007/s11904-012-0115-y. PMID 22415474
- [Background] Cohen J. The emerging race to cure HIV infections. Science. 2011 May 13;332(6031):784-5, 787-9. doi: 10.1126/science.332.6031.784. No abstract available. PMID 21566173
- [Background] Lewin SR, Evans VA, Elliott JH, Spire B, Chomont N. Finding a cure for HIV: will it ever be achievable? J Int AIDS Soc. 2011 Jan 24;14:4. doi: 10.1186/1758-2652-14-4. PMID 21255462
- [Derived] Katlama C, Lambert-Niclot S, Assoumou L, Papagno L, Lecardonnel F, Zoorob R, Tambussi G, Clotet B, Youle M, Achenbach CJ, Murphy RL, Calvez V, Costagliola D, Autran B; EraMune-01 study team. Treatment intensification followed by interleukin-7 reactivates HIV without reducing total HIV DNA: a randomized trial. AIDS. 2016 Jan;30(2):221-30. doi: 10.1097/QAD.0000000000000894. PMID 26684819